CLINICAL TRIAL: NCT01040208
Title: Safety of Flibanserin Versus Placebo in Women Taking a Selective Serotonin Reuptake Inhibitor or Norepinephrine Serotonin Reuptake Inhibitor With Decreased Sexual Desire
Brief Title: 12 Week Safety Trial of Flibanserin in Depressed Women Taking an SSRI or SNRI With Decreased Sexual Desire and Distress
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by Sponsor for administrative reasons prior to completion
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 511.114
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-07

CONDITIONS: Sexual Dysfunctions, Psychological; Depression
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Depression | interventions — flibanserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- flibanserin 50 mg to 100 mg qhs (Experimental): Patient to receive one tablet of flibanserin 50 mg and one tablet of flibanserin placebo qhs for 14 days then will receive 2 flibanserin tablets of 50 mg qhs
  Interventions: Drug: flibanserin 50 mg to 100 mg qhs
- flibanserin 100 mg qhs (Experimental): Patient to receive 2 flibanserin tablets of 50 mg qhs
  Interventions: Drug: flibanserin 100 mg qhs
- placebo 2 tablets qhs (Experimental): Patient to receive 2 placebo tablets of 50 mg qhs
  Interventions: Drug: placebo 2 tablets qhs

INTERVENTIONS:
Drug: flibanserin 50 mg to 100 mg qhs — 50 to 100mg qhs
  Arms: flibanserin 50 mg to 100 mg qhs
Drug: flibanserin 100 mg qhs — 100mg qhs
  Arms: flibanserin 100 mg qhs
Drug: placebo 2 tablets qhs — 50 mg placebo
  Arms: placebo 2 tablets qhs

SUMMARY:
The current trial will explore the safety of flibanserin in combination with Selective Serotonin Reuptake Inhibitors or Norepinephrine Serotonin Reuptake Inhibitors in a representative population of women with depressive and possible concurrent anxiety symptomatology.

ELIGIBILITY:
Inclusion criteria:

1. Women 18-50 years of age, not postmenopausal at the Screen Visit
2. Women with mild/remitted depressive disorder with score of <11 on the Quick Inventory of Depressive Symptoms Self Report and <16 on the Beck Anxiety Inventory at Screen/Baseline Visits
3. Women with decreased sexual desire and distress present at least 4 weeks at Screen Visit as determined by the Clinical Interview for Female Sexual Dysfunction-Depression and Diagnostic and Statistical Manual IV-Text Revision (DSM IV-TR)
4. Score of 15 or higher on the Female Sexual Distress Scale-Revised at Screen/Baseline Visits
5. Score of 9 or lower on the Changes in Sexual Functioning Questionnaire-Female desire/interest item at Screen/Baseline Visits
6. Patients must be taking the same Selective Serotonin Reuptake Inhibitor or Norepinephrine Serotonin Reuptake Inhibitor for 3 months and be on a stable dose at least 2 months before the Screen Visit and remain on this regimen during the trial and for 1 month after trial completion
7. Patients must have had no treatment for Female Sexual Dysfunction 2 months before Screen Visit
8. Patients must use medically accepted contraception method
9. Patients must be in a secure, stable, monogamous, heterosexual relationship at least 12 months prior to Screen Visit, according to the Clinical Interview for Female Sexual Dysfunction-Depression

Exclusion criteria:

Conditions which may interfere with the ability to participate include, but are not limited to:

1. Patients who have taken any Prohibited Medications within 30 days before Baseline Visit
2. Patients with history of drug dependence/abuse (including alcohol) within past year
3. Patients with history of participation in a trial of another investigational drug within 1 month prior to the Screen Visit, or participation in previous flibanserin study
4. Women with lifelong decreased sexual desire (or Hypoactive Sexual Desire Disorder), Female Sexual Arousal Disorder and/or Female Orgasmic Disorder, per DSM IV-TR criteria
5. Patients who meet DSM IV-TR criteria for Sexual Aversion Disorder, Substance-Induced Sexual Dysfunction other than Selective Serotonin Reuptake Inhibitor/Norepinephrine Serotonin Reuptake Inhibitor-Induced Sexual Dysfunction, Dyspareunia, Vaginismus, Gender Identity Disorder, Paraphilia, or Sexual Dysfunction Due to a General Medical Condition
6. Patients who have had a hysterectomy, or are in the post menopause stage (i.e., bilateral oophorectomy, chemically induced menopause)
7. Patients with history of pelvic inflammatory disease, urinary tract, vaginal infection/vaginitis, cervicitis, interstitial cystitis, vulvodynia, significant vaginal atrophy in the 4 weeks before the Screen Visit
8. Patients who are breastfeeding or have breastfed within 6 months prior to the Baseline Visit.
9. Patients who are pregnant (by serum pregnancy test) or have been pregnant within 6 months prior to the Baseline Visit
10. Patients with current Depressive Disorder (may have concurrent mild Anxiety Disorder) not adequately controlled during the last 2 months and/or with a score of <11 on the Quick Inventory of Depressive Symptoms Self Report and/or a score of <16 on the Beck Anxiety Inventory at Screen and/or Baseline Visits
11. Patients with history of suicide attempt within the last year or current suicidal ideation. Investigator must assess history of suicidality to determine if patient is at risk before entering the trial
12. Patients with history of other psychiatric disorders that could impact sexual function, risks patient safety, or may impact compliance. Axis I disorders (except anxiety symptoms and disorders) are excluded. Axis II disorders are allowed
13. Patients with significant cardiac, neurologic, hepatic, renal, hematologic, respiratory, gastrointestinal, immunological, endocrine disease
14. Patients with history of breast cancer or other cancer within the last 5 years, other than non-invasive, previously resected skin cancer

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (42):
- United States (42):
  - Clinical Innovations, Costa Mesa, California
  - Mood & Anxiety Research, Fresno, California
  - Synergy Clinical Research Center, National City, California
  - Clinical Innovations, Riverside, California
  - Schuster Medical Research, Sherman Oaks, California
  - Diablo Clinical Research, Walnut Creek, California
  - Western Affiliated Research Institute, Denver, Colorado
  - Radiant Research, Denver, Colorado
  - Ali Kashfi, Altamonte Springs, Florida
  - Gulf Coast Clinical Research, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Kolin Research Group, Winter Park, Florida
  - Atlanta Institute of Medicine & Research, Atlanta, Georgia
  - Comprehensive Neuroscience, Atlanta, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Capstone Clinical Research, Livertyville, Illinois
  - Psychiatric Medicine Associates, Skokie, Illinois
  - Clinco, Terre Haute, Indiana
  - Clinical Trials Technology, Prairie Village, Kansas
  - Sheppard Pratt Hospital, Baltimore, Maryland
  - ActivMed Practices and Research, Haverhill, Massachusetts
  - Millennium Psychiatric Associates, Creve Coeur, Missouri
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Neurobehavioral Research, Cedarhurst, New York
  - Bioscience Research, Mount Kisco, New York
  - Medical and Behavioral Health Research, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - MIdwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Future Search Trials, Austin, Texas
  - Mary Ann Knesevich, Irving, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - San Antonio Psychiatric Research Center, San Antonio, Texas
  - Alliance Research Group, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Flibanserin 50 mg to 100 mg Qhs (Take Daily, at Bedtime): Patient to receive one tablet of flibanserin 50 mg and one tablet of flibanserin placebo qhs for 14 days then will receive 2 flibanserin tablets of 50 mg qhs
- Placebo 2 Tablets Qhs: Patient to receive 2 flibanserin placebo tablets of 50 mg qhs
Period: Overall Study
Arm/Group | Flibanserin 50 mg to 100 mg Qhs (Take Daily, at Bedtime) | Flibanserin 100 mg Qhs | Placebo 2 Tablets Qhs
Started | 45 | 28 | 38
Completed | 39 | 15 | 35
Not Completed | 6 | 13 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flibanserin 50 mg to 100 mg Qhs | Flibanserin 100 mg Qhs | Placebo 2 Tablets Qhs | Total
Number analyzed (Participants) | 45 | 28 | 38 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 28 | 38 | 111
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (7.2) | 36.9 (8.0) | 37.7 (7.1) | 37.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 28 | 38 | 111
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 28 | 38 | 111

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint is the Occurrence of Adverse Events During the Treatment and Post Treatment Period.
Time Frame: 17 weeks
Population: The treated set (TS) consisted of those patients who were dispensed study medication and who were documented to have taken at least one dose of study medication. All analyses were conducted on the TS.
Measure: Number; unit: participants
Arm/Group | Flibanserin 50 mg to 100 mg Qhs | Flibanserin 100 mg Qhs | Placebo 2 Tablets Qhs
Number analyzed (Participants) | 45 | 28 | 38
participants | 16 | 14 | 32

2. Secondary Outcome: The Occurrence of Mild Depressive Symptoms (i.e., a Total Score of '7' to '11', Inclusive) That Have Remitted (i.e., a Total Score of '6' or Less) on the 16 Item Quick Inventory of Depressive Symptoms - Self Report at Visit 6 (Week 12)
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Flibanserin 50 mg to 100 mg Qhs | Flibanserin 100 mg Qhs | Placebo 2 Tablets Qhs
Number analyzed (Participants) | 45 | 28 | 38
participants | 8 | 6 | 4

3. Secondary Outcome: The Occurrence of Mild Anxiety Symptoms (i.e., a Total Score of '8' to '16', Inclusive) That Have Remitted (i.e., a Total Score of '7' or Less) on the Beck Anxiety Inventory at Visit 6 (Week 12)
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Flibanserin 50mg to 100mg Qhs: Group includes the 45 patients who took flibanserin 50 mg q.h.s. for the first 2 weeks followed by flibanserin 100 mg q.h.s.
Arm/Group | Flibanserin 50mg to 100mg Qhs | Flibanserin 100mg Qhs | Placebo 2 Tablets Qhs
Number analyzed (Participants) | 45 | 28 | 38
participants | 8 | 4 | 1

ADVERSE EVENTS:
Arm/Group | Flibanserin 50 mg to 100 mg Qhs | Flibanserin 100 mg Qhs | Placebo 2 Tablets Qhs
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/28 | 0/38
Other Adverse Events (participants affected / at risk) | 16/45 | 14/28 | 32/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 50 mg to 100 mg Qhs (N=45) | Flibanserin 100 mg Qhs (N=28) | Placebo 2 Tablets Qhs (N=38)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 7 (7)
Sedation (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1) | 2 (2)
Weight increased (Investigations) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No